CLINICAL TRIAL: NCT06549374
Title: Kinetics of INF-γ Production in Intensive Care Patients-Monitoring of INF-γ in Intensive Care
Brief Title: Kinetics of INF-γ Production in Intensive Care Patients
Acronym: IGREY
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240860
Record Dates: First submitted 2024-07-29; First posted 2024-08-12 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-04

CONDITIONS: Intensive Care
Keywords: INF-γ; Inflammation; immunostimulation
MeSH Terms: conditions — Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults in Intensive care: Patient included will be adult patients admitted to intensive care after severe trauma, high-risk surgery, or presenting with acute respiratory distress
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — After informing eligible patients (or their trusted support person, relative/guardian/curator where applicable) and in the absence of any opposition, they are included in the research.
  Blood samples from an arterial catheter already in place will be taken every day from D1 to D7, then every 72 hours until discharge from intensive care, or until D28. For each of these samples, a maximum volume of 4 ml will be collected in a heparinized tube. Samples will not be taken if the hemoglobin level is below 7g/dl. For patients undergoing controlled surgery, the D1 sample will be taken as soon as possible after induction of anaesthesia.
  Patients will be monitored until discharge from intensive care, or until D28 at the latest. Apart from the blood samples included in this study, all other examinations will be carried out as part of routine management. Data will be collected exclusively from medical records.

SUMMARY:
Most patients admitted to intensive care after severe trauma, high-risk surgery, or acute respiratory distress are frequently characterized by significant initial inflammation accompanied by a compensatory anti-inflammatory response, which can lead to profound post-aggressive immunosuppression. This immunosuppression is associated with an increased risk of nosocomial infections, viral reactivations, prolonged ICU stays, and ultimately, increased mortality. Consequently, immunostimulation with agents such as interferon gamma (IFN-γ) has been proposed as a means to restore immune defense in the most severe patients. However, in a recent study conducted on mechanically ventilated patients with acute organ failure, treatment with interferon gamma-1b compared to placebo did not significantly reduce the incidence of nosocomial pneumonia or 28-day mortality and was even associated with an increase in severe side effects, leading to the premature termination of the trial. These results, along with previous studies, suggest that for IFN-γ to be effective, it must be targeted at patients who have reached the immunosuppressive phase. In the absence of evident clinical signs, the use of biomarkers could guide clinicians in identifying the appropriate patients and the optimal timing for this therapy.

In a recent monocentric study, they evaluated a new automated IFN-γ assay on a cohort of 22 septic patients to monitor T lymphocyte functionality independently of antigen. As expected, the results showed a marked decrease in IFN-γ release, which correlated with altered classical cellular parameters (CD8+ T cells, mHLA-DR). Since the test is performed using whole blood, requires no technician intervention, and provides results within four hours, this project propose to characterize the evolution of the immune status of a large cohort of ICU patients, including those with severe trauma, high-risk surgery, or acute respiratory distress syndrome.

DETAILED DESCRIPTION:
Most patients admitted to intensive care after severe trauma, high-risk surgery, or acute respiratory distress are frequently characterized by significant initial inflammation accompanied by a compensatory anti-inflammatory response, which can lead to profound post-aggressive immunosuppression. This immunosuppression is associated with an increased risk of nosocomial infections, viral reactivations, prolonged ICU stays, and ultimately, increased mortality. Consequently, immunostimulation with agents such as interferon gamma (IFN-γ) has been proposed as a means to restore immune defense in the most severe patients. However, in a recent study conducted on mechanically ventilated patients with acute organ failure, treatment with interferon gamma-1b compared to placebo did not significantly reduce the incidence of nosocomial pneumonia or 28-day mortality and was even associated with an increase in severe side effects, leading to the premature termination of the trial. These results, along with previous studies, suggest that for IFN-γ to be effective, it must be targeted at patients who have reached the immunosuppressive phase. In the absence of evident clinical signs, the use of biomarkers could guide clinicians in identifying the appropriate patients and the optimal timing for this therapy.

Among the described immune alterations and associated biomarkers in critically ill patients, the decrease in Human Leukocyte Antigen (HLA-DR) expression on monocytes (mHLA-DR) has been studied more extensively and is now considered a reliable biomarker for guiding myeloid-targeted immunotherapies. While functional tests are the best means to explore acquired immunosuppression in the ICU, as they directly measure the capacity of a given cell population to respond to an in vitro stimulus, they present analytical obstacles to their deployment. Most protocols are "homemade" and lack standardization, which is a major obstacle to large-scale trials and their use in clinical practice.

In a recent monocentric study, they evaluated a new automated IFN-γ assay on a cohort of 22 septic patients to monitor T lymphocyte functionality independently of antigen. As expected, the results showed a marked decrease in IFN-γ release, which correlated with altered classical cellular parameters (CD8+ T cells, mHLA-DR). Since the test is performed using whole blood, requires no technician intervention, and provides results within four hours, this project propose to characterize the evolution of the immune status of a large cohort of ICU patients, including those with severe trauma, high-risk surgery, or acute respiratory distress syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Patients admitted to intensive care after severe trauma, or presenting with acute respiratory distress, or undergoing cardiac, vascular, or digestive surgery with planned postoperative intensive care. Exclusion Criteria

Exclusion Criteria:

* Expressed opposition from the patient, a relative (if applicable), or their legal representative (guardian, curator)
* Pregnant woman
* Hemoglobin less than 7g/dl at inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient included will be adult patients admitted to intensive care after severe trauma, high-risk surgery, or presenting with acute respiratory distress
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2026-04-24 (Estimated); Study Completion 2026-05-24 (Estimated)

PRIMARY OUTCOMES:
INF-γ production in patients admitted to intensive care after severe trauma, high-risk surgery, or acute respiratory distress | Daily value from day 1 to day 7, then every 72 hours until discharge from intensive care (assessed up to day 28).
  The measurement of INF-γ production will be conducted using a fully automated Interferon Gamma Realease Assay (IGRA) test.

SECONDARY OUTCOMES:
ICU discharge Vital status | at ICU discharge, and at the latest Day 28
  Vital status at discharge from ICU
Incidence of nosocomial infections | From ICU-admission to ICU-discharge, and at the latest Day 28
  Incidence of nosocomial infections occurring in the ICU : number, type, and duration of antibiotic therapy
Incidence of viral reactivations for CMV and HSV | From ICU-admission to ICU-discharge, and at the latest Day 28
  Incidence of viral reactivations as detected by PCR for CMV (Cytomegalovirus) and HSV (Herpes Simplex Virus) in the ICU
Length of mechanical ventilation | From ICU-admission to ICU-discharge, and at the latest Day 28
  Duration of mechanical ventilation in ICU
Presence of septic shock | From ICU-admission to ICU-discharge, and at the latest Day 28
  Presence of septic shock in the ICU
Renal impairment | From ICU-admission to ICU-discharge, and at the latest Day 28
  Renal impairment defined by a Kidney Disease Improving Global Outcomes (KDIGO) score > 1.
  Scale of 1 to 3, with 3 corresponding to severe acute kidney damage.
mHLA-DR expression | Daily value from day 1 to day 7, then every 72 hours until discharge from intensive care (assessed up to day 28).
  mHLA-DR expression by flow cytometry
Length of ICU stay | at ICU discharge, and at the latest day 28
  Length of stay in intensive care

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Reanimation department, Annecy Genevois hospital, Annecy
  - Reanimation department, Clermont-Ferrand Hospital, Clermont-Ferrand
  - Reanimation department, Lyon hospital, Lyon
  - Réanimation cardio-chirurgicale - Pitié-Salpêtrière hospital, Paris, Île-de-France Region
  - Réanimation chirurgicale Gaston Cordier - Pitié-Salpêtrière hospital, Paris, Île-de-France Region
  - Réanimation chirurgicale Husson Mourrier - Pitié-Salpêtrière hospital, Paris, Île-de-France Region
  - Réanimation neuro-chirurgicale - Pitié-Salpêtrière hospital, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor.
Access Criteria: Researchers who provide a methodologically sound proposal.